CLINICAL TRIAL: NCT06409845
Title: Effectiveness and Tolerability of Eptinezumab: a Prospective, Multicentric, Cohort Study
Brief Title: Effectiveness and Tolerability of Eptinezumab
Acronym: TACHIS
Status: Recruiting | Type: Observational
Sponsor: University of Florence (Other)
Collaborators: Azienda Ospedaliero Universitaria Policlinico Modena (Other); Società Italiana per lo Studio delle Cefalee (Other); IRCCS National Neurological Institute "C. Mondino" Foundation (Other); Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other); Università degli Studi dell'Aquila (Other); University of Roma La Sapienza (Other); Euganea Health Unit, Padua, Italy (Unknown); Azienda Ospedaliero-Universitaria di Parma (Other); Azienda Ospedaliera S. Maria della Misericordia (Other); A.O.U. Città della Salute e della Scienza (Other); Cliniche Humanitas Gavazzeni (Other); University of Campania Luigi Vanvitelli (Other); Ospedale Santo Stefano (Other); Azienda Policlinico Umberto I (Other); Auxologico San Luca (Other); Asst Degli Spedali Civili Di Brescia (Other); Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Principal Investigator, Luigi Francesco Iannone, Researcher at the Headache Center and Clinical Pharmacology Unit and the Department of Health Sciences, University of Florence, Principal Investigator, University of Florence
Other Study IDs: RICe_5
Record Dates: First submitted 2024-04-05; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Migraine; Migraine With Aura; Migraine Without Aura; Chronic Migraine
Keywords: Headache; Medication overuse headache; Pain; Migraine prevention; Anti-CGRP monoclonal antibodies; eptinezumab
MeSH Terms: conditions — Migraine Disorders; Migraine with Aura; Migraine without Aura; Headache; Headache Disorders, Secondary; Pain | interventions — eptinezumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Episodic migraine: Patients affected by migraine with an episodic pattern (< 15 monthly migraine days) with or without aura according to ICHD-III criteria.
  Interventions: Drug: Eptinezumab 100 or 300 mg ev
- Chronic migraine: atients affected by chronic migraine (> 15 monthly headache days with at least 8 days with migraine features) according to ICHD-III criteria.
  Interventions: Drug: Eptinezumab 100 or 300 mg ev

INTERVENTIONS:
Drug: Eptinezumab 100 or 300 mg ev — Patients administered eptinezumab 100 or 300 mg ev quarterly for migraine prevention
  Other Names: Eptinezumab

SUMMARY:
The purpose of this prospective and multicentric study is to evaluate the effectiveness and tolerability of eptinezumab as preventive migraine treatment in a cohort of episodic or chronic migraine patients.

DETAILED DESCRIPTION:
Eptinezumab belongs to the monoclonal antibodies directed against the calcitoning gene related peptide - CGRP (mAbs). It is actually the only mAb administered intravenously, currently available at the dose of 100 or 300mg with a quarterly iv infusion.

It has an indication for migraine prevention for episodic and chronic migraine. Previous randomized, placebo-controlled clinical trials proved its effectiveness in the preventive setting for patients with episodic and chronic migraine.

Moreover, a previous study also supported evidence of faster headache pain freedom and most bothersome symptom resolution after eptinezumab 100mg infusion during migraine acute attack compared to placebo.

RCTs also demonstrated a good tolerability profile. The most commonly reported adverse events were mainly upper respiratory tract infections, fatigue and hypersensitivity reactions.

In this prospective multicentric study the investigators aim to evaluate eptinezumab effectiveness and tolerability as preventive migraine treatment in a real-world setting.

Subjects who meet the inclusion criteria will be enrolled and will participate in the study. Baseline demographic and clinical data will be collected at the baseline visit. The observation period will last for two years during which patients will be administered eptinezumab 100 or 300 mg according to clinicians' judgment, for a time period related to Italian Medicines Agency reimbursability criteria.

Data will be collected at baseline and every three months, up to two years. Subjects will be asked to keep a headache diary to collect monthly headache and migraine days, migraine severity, associated symptoms and drug consumption. Questionnaires will be collected every three months.

Data collection will focus on: i) demographic data, ii) migraine history, iii) pain intensity, iv) presence and evolution of migraine associated symptoms and aura, v) migraine associated disability, vi) tolerability and eventual treatment- emergent adverse events, vii) treatment persistence, viii) questionnaires related to disability, allodynia, quality of life, interictal burden and effectiveness of the ongoing acute and preventive treatments. The online database REDCap will be used for data collection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine without aura, migraine with aura, or chronic migraine according to the 3rd edition of the International Classification of Headache Disorder (ICHD-III);
* Good compliance to study procedures;
* Availability of headache diary at least of the preceding months before enrolment;
* At least 8 monthly migraine days.

Exclusion Criteria:

* Subjects with contraindications for use of eptinezumab;
* Concomitant diagnosis of medical diseases and/or comorbidities that, in the Investigator's opinion might interfere with study assessments;
* medical comorbidities that could interfere with study results;
* Pregnancy and breastfeeding
* Changes in preventive treatments in the month before the first administration of eptinezumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multicentric study on patients attending the outpatient clinic of Italian Headache centres who meet criteria for eptinezumab use as migraine preventive treatment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Changes in migraine frequency after three months of treatment | Baseline (T0) - 3 months of treatment with eptinezumab (T3)
  Changes in monthly migraine days after three months of treatment with eptinezumab compared to baseline (continuous variable)
Percentage of 50% Responders (namely patients who presented a reduction of MMDs >/ = 50% compared to baseline) after three months of treatment | Baseline (T0) - 3 months of treatment with eptinezumab (T3)
  Percentage of 50% Responders (namely patients who presented a reduction of MMDs >/ = 50% compared to baseline) after three months of treatment with eptinezumab (continuous variable)

SECONDARY OUTCOMES:
Changes in migraine frequency across twelve months of eptinezumab treatment | Baseline (T0) - 6 months (T6) - 12 months (T12) of treatment with eptinezumab
  Changes in monthly migraine days after six and twelve months of treatment with eptinezumab compared to baseline (continuous variable)
Percentage of 50% Responders (namely patients who presented a reduction of MMDs >/ = 50% compared to baseline) across twelve months of treatment with eptinezumab | Baseline (T0) - 6 months (T6) - 12 months (T12) of treatment with eptinezumab
  Percentage of 50% Responders (namely patients who presented a reduction of MMDs >/ = 50% compared to baseline) after six and twelve months of treatment with eptinezumab (continuous variable)
Evaluation of any adverse event (qualitative) | 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with eptinezumab
  Type of any adverse events in patients receiving eptinezumab during the observation period (categorical variable)
Evaluation of any adverse event (quantitative) | 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with eptinezumab
  Percentage of reported adverse events in patients receiving eptinezumab assessed quarterly during the observation period (continuous variable)
Evaluation of serious adverse events | 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with eptinezumab
  Percentage of serious adverse events (namely those resulting in death, is life-threatening, requires hospitalisation or prolongation of existing hospitalisation, results in persistent or significant disability or incapacity, or is a birth defect) in patients receiving eptinezumab during the observation period (continuous variable)
Evaluation of adverse events leading to treatment discontinuation | 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with eptinezumab
  Percentage of adverse events leading to treatment discontinuation in patients receiving eptinezumab during the observation period (continuous variable)
Consistency of treatment response | 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with eptinezumab
  Percentage of patients with a stable 50% response across twelve months of eptinezumab treatment (continuous variable)
Changes in migraine disability (MIDAS) | 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with eptinezumab
  Changes in MIgraine Disability ASsesment questionnaire across treatment (continuous variable, 0-270 scale, higher scores indicate higher disability: 0-5, little/no disability; 6-10, mild disability; 11-20, moderate disability; >20, severe disability)
Changes in migraine disability (HIT-6) | 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with eptinezumab
  Changes in Headache Impact Test-6 questionnaire across treatment (continuous variable, 36-78 scale, higher scores indicates greater disability)
Changes in response to acute migraine treatment (m-TOQ) | 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with eptinezumab
  Changes in migraine Treatment Optimization Questionnaire across eptinezumab treatment (continuous variable, 0-8 scale, higher score indicates higher acute therapy effectiveness)
Changes in allodynia (ASC-12) | 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with eptinezumab
  Changes in Allodynia Symptoms Checklist-12 questionnaire across treatment (continuous variable, 0-24 scale, higher score indicates more severe allodynia)
Changes in interictal burden across eptinezumab treatment (MIBS-4) | 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with eptinezumab
  Changes in Migraine Interictal Burden Scale-4 questionnaire across treatment (continuous variable, 0-4 scale, 0 indicates no interictal burden, 1-2 mild level of interictal burden, 3 moderate interictal burden, 4 severe interictal burden)
Percentage of patients with Medication overuse headache reverted during treatment | 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with eptinezumab
  Percentage of patients with a baseline diagnosis of MOH reverted after 3 - 6 and 12 months of eptinezumab treatment (continuous variable)

OTHER OUTCOMES:
Changes in the number of monthly migraine days with aura (quantitative) | 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with eptinezumab
  Changes in monthly migraine days with aura across twelve months treatment (continuous variable)
Variation of duration of aura (qualitative) | 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with eptinezumab
  Changes in duration of aura across eptinezumab treatment (categorical variable - minutes, assessed through headache diary)
Variation of type of aura (qualitative) | 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with eptinezumab
  Changes in type of aura across eptinezumab treatment (assessed through headache diary and anamnestic data collection)
MMDs reduction in patients Non-responders to other anti-CGRP mAbs | 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with eptinezumab
  Change of monthly migraine days across eptinezumab twelve-months treatment in those patients who did not respond to other anti-CGRP mAbs (continuous variable)
Percentage of 50% Responders in patients Non-responders to other anti-CGRP mAbs | 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with eptinezumab
  Percentage of 50% Responders across eptinezumab treatment in those patients who did not respond to anti-CGRP mAbs (continuous variable)
Changes in migraine duration across treatment | 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with eptinezumab
  Changes in migraine duration (continuous variable, hours, assessed through a paper diary)
Changes in migraine severity across treatment | 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with eptinezumab
  Changes in migraine severity across treatment (continuous variable, 0-10 numerical rating scale, higher scores indicate higher severity)
Changes in duration of the most bothersome symptom(s) | 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with eptinezumab
  Changes in duration of the most bothersome symptom(s) across treatment (continuous variable: minutes, assessed through a paper diary)
Changes in severity of the most bothersome symptom(s) | 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with eptinezumab
  Changes in durantion and severity of the most bothersome symptom(s) (continuous variable: 0-10 numerical rating scale, higher scores indicate higher severity)
Changes in self-reported effectiveness of eptinezumab treatment | 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with eptinezumab
  Changes in Patients Global Impression of Change (PGIC) questionnaire across treatment (continuous variable)
Changes in self-reported effectiveness of acute treatment | 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with eptinezumab
  Changes in self-reported effectiveness of usual acute treatment (qualitative variable)
Changes in perimenstrual attacks | 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with eptinezumab
  Changes in duration, intensity and associated symptoms of perimenstrual attacks

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - SOD Centro Cefalee e Farmacologia Clinica, AOU Careggi, Florence
  - AOU Policlinico Di Modena, Modena

REFERENCES:
- [Background] Dodick DW, Lipton RB, Silberstein S, Goadsby PJ, Biondi D, Hirman J, Cady R, Smith J. Eptinezumab for prevention of chronic migraine: A randomized phase 2b clinical trial. Cephalalgia. 2019 Aug;39(9):1075-1085. doi: 10.1177/0333102419858355. Epub 2019 Jun 24. PMID 31234642
- [Background] Winner PK, McAllister P, Chakhava G, Ailani J, Ettrup A, Krog Josiassen M, Lindsten A, Mehta L, Cady R. Effects of Intravenous Eptinezumab vs Placebo on Headache Pain and Most Bothersome Symptom When Initiated During a Migraine Attack: A Randomized Clinical Trial. JAMA. 2021 Jun 15;325(23):2348-2356. doi: 10.1001/jama.2021.7665. PMID 34128999
- [Background] Ashina M, Lanteri-Minet M, Pozo-Rosich P, Ettrup A, Christoffersen CL, Josiassen MK, Phul R, Sperling B. Safety and efficacy of eptinezumab for migraine prevention in patients with two-to-four previous preventive treatment failures (DELIVER): a multi-arm, randomised, double-blind, placebo-controlled, phase 3b trial. Lancet Neurol. 2022 Jul;21(7):597-607. doi: 10.1016/S1474-4422(22)00185-5. PMID 35716692